CLINICAL TRIAL: NCT01366534
Title: Safety, Immunogenicity and Efficacy Against Malaria in the Sporozoite Challenge Model of One Dose of Ad35.CS.01 Malaria Vaccine Followed by Two Doses of Malaria 257049 Vaccine in Healthy Malaria-naïve Adults
Brief Title: Safety, Immunogenicity and Efficacy Against of a Combined Malaria Vaccine in Healthy Malaria-naïve Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: The PATH Malaria Vaccine Initiative (MVI) (Other); Crucell Holland BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 114460
Record Dates: First submitted 2011-06-02; First posted 2011-06-06 (Estimated); Results first posted 2017-06-09 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Malaria
Keywords: safety; Vaccine; Phase 1/2; immunogenicity; Malaria; efficacy; sporozoite challenge
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- Ad35.CS.01 Group (Experimental): Healthy male or non-pregnant female subjects, aged 18 to 50 years, were administered one dose of Ad35.CS.01 vaccine at Month 0, and 2 doses of GSK257049 at Months 1 and 2 intramuscularly in the deltoid of the non-dominant arm. The duration of the study was approximately 11 months for vaccinated subjects.
  Interventions: Biological: Crucell's replication deficient adenovirus type 35 circumsporozoite malaria vaccine (Ad35.CS.01); Biological: GSK Biologicals' malaria vaccine 257049 (2 doses)
- GSK257049 Group (Experimental): Healthy male or non-pregnant female subjects, aged 18 to 50 years, were administered 3 doses of GSK257049 vaccine at Months 0, 1 and 2 intramuscularly in the deltoid of the non-dominant arm. The duration of the study was approximately 11 months for vaccinated subjects.
  Interventions: Biological: GSK Biologicals' malaria vaccine 257049 (3 doses)
- Control Group (Experimental): Healthy male or non-pregnant female subjects, aged 18 to 50 years, were volunteers who did not receive any immunization but were subjected to the sporozoite challenge. The duration of the study was approximately 8 months for infectivity control subjects.
  Interventions: Other: Sporozoite challenge

INTERVENTIONS:
Biological: Crucell's replication deficient adenovirus type 35 circumsporozoite malaria vaccine (Ad35.CS.01) — One dose will be administered intramuscularly at Study Day 0.
  Arms: Ad35.CS.01 Group
Biological: GSK Biologicals' malaria vaccine 257049 (2 doses) — Two doses will be administered intramuscularly at monthly intervals
  Arms: Ad35.CS.01 Group
Biological: GSK Biologicals' malaria vaccine 257049 (3 doses) — Three doses will be administered intramuscularly at monthly intervals
  Arms: GSK257049 Group
Other: Sporozoite challenge — Subjects were challenged with sporozoite-infected mosquitoes to determine whether immune protective response had been induced by vaccination.
  Arms: Control Group

SUMMARY:
This study will evaluate whether administration of two investigational malaria vaccines (257049 and Ad35.CS.01 vaccines) combined in one immunization schedule increases protection against malaria infection as compared to protection induced by the 257049 vaccine alone. The study will also evaluate the safety and the immune response to the new combination of the two experimental malaria vaccines.

DETAILED DESCRIPTION:
Approximately 168 healthy, malaria-naïve volunteers aged 18 - 50 years, divided into 2 groups (84 in each group), will receive either one dose of Ad35.CS.01 followed by two doses of 257049 at monthly intervals or 3 doses of 257049 vaccine at monthly intervals. Of these, a maximum of 138 vaccinated volunteers will be challenged with P. falciparum infected mosquitoes. The challenge will occur 2 weeks following the third immunization. A group of up to 18 infectivity controls will begin participation in the study at the challenge stage. These controls receive no vaccine and are enrolled for malaria-challenge only in order to provide comparison group for vaccinated individuals.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes can and will comply with the requirements of the protocol.
* A male or non-pregnant female 18 to 50 years of age at the time of first vaccination.
* Written informed consent obtained from the subject before screening procedures.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.
* Available to participate for the duration of the study.
* Female subjects of non-childbearing potential.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate Food and Drug Administration (FDA)-approved contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination, and
  * has agreed to continue adequate FDA-approved contraception during the entire treatment period and for 2 months after completion of the vaccination series and/or malaria challenge.
* Pass a comprehension assessment test.

Exclusion Criteria:

* Use of any investigational or non-registered product within 30 days preceding the first dose of study vaccine, or planned use of any investigational or non-registered product other than the study vaccines during the study period.
* Planned administration/ administration of a vaccine not foreseen by the study protocol within 7 days of the first dose of vaccines.
* Prior receipt of an investigational malaria or adenovirus vaccine.
* Chronic use of antibiotics with antimalarial effects.
* History of malaria chemoprophylaxis within 60 days prior to vaccination.
* Any history of malaria.
* Planned travel to malaria endemic areas during the study period.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine(s) including latex.
* History of allergic disease or reactions likely to be exacerbated by chloroquine.
* History of psoriasis and porphyria, which may be exacerbated after chloroquine treatment.
* Current use of medications known to cause drug reactions to chloroquine, such as antacids and kaolin.
* Any history of anaphylaxis in reaction to any previous vaccination.
* History of severe reactions to mosquito bites.
* Administration of immunoglobulins and/or any blood products within the three months preceding the first dose of study vaccine or planned administration during the study period.
* Chronic administration of immunosuppressants or other immune modifying drugs within six months prior to first vaccine dose.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including immunodeficiency virus (HIV) infection.
* Family history of congenital or hereditary immunodeficiency.
* History of splenectomy.
* Major congenital defects or serious chronic illness.
* History of any neurological disorders or seizures.
* Acute disease and/or fever at the time of enrollment.
* Acute disease is defined as the presence of a moderate or severe illness with or without fever. Subjects with a minor illness without fever may be enrolled at the discretion of the investigator.
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests.
* Any abnormal baseline laboratory screening tests.
* Evidence of increased cardiovascular disease risk, "moderate" or "high", according to the NHANES I criteria.
* An abnormal baseline screening electrocardiogram (EKG).
* Hepatomegaly, right upper quadrant abdominal pain or tenderness.
* Personal history of autoimmune disease.
* Seropositive for hepatitis B surface antigen or Hepatitis C virus (antibodies to HCV).
* Pregnant or lactating female.
* Female who intends to become pregnant during the study or planning to discontinue contraceptive measures.
* Suspected or known current alcohol abuse.
* Chronic or active intravenous drug use.
* History of blood donation within 56 days preceding enrolment.
* Any other significant finding that in the opinion of the investigator would increase the risk of having an adverse outcome from participating in this study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2011-08-10 (Actual); Primary Completion 2012-02-27 (Actual); Study Completion 2012-07-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Silver Spring, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study is available via the Clinical Study Data Request site (click on the link provided below)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Patient-level data for this study is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Background] Ockenhouse CF, Regules J, Tosh D, Cowden J, Kathcart A, Cummings J, Paolino K, Moon J, Komisar J, Kamau E, Oliver T, Chhoeu A, Murphy J, Lyke K, Laurens M, Birkett A, Lee C, Weltzin R, Wille-Reece U, Sedegah M, Hendriks J, Versteege I, Pau MG, Sadoff J, Vanloubbeeck Y, Lievens M, Heerwegh D, Moris P, Guerra Mendoza Y, Jongert E, Cohen J, Voss G, Ballou WR, Vekemans J. Ad35.CS.01-RTS,S/AS01 Heterologous Prime Boost Vaccine Efficacy against Sporozoite Challenge in Healthy Malaria-Naive Adults. PLoS One. 2015 Jul 6;10(7):e0131571. doi: 10.1371/journal.pone.0131571. eCollection 2015. PMID 26148007
- [Derived] Spreng RL, Seaton KE, Lin L, Hilliard S, Horn GQ, Abraha M, Deal AW, Li K, Carnacchi AJ, Feeney E, Shabbir S, Zhang L, Bekker V, Mudrak SV, Dutta S, Mercer LD, Gregory S, King CR, Wille-Reece U, Jongert E, Kisalu NK, Tomaras GD, Dennison SM. Identification of RTS,S/AS01 vaccine-induced humoral biomarkers predictive of protection against controlled human malaria infection. JCI Insight. 2024 Oct 8;9(19):e178801. doi: 10.1172/jci.insight.178801. PMID 39377226
- [Derived] Li K, Dodds M, Spreng RL, Abraha M, Huntwork RHC, Dahora LC, Nyanhete T, Dutta S, Wille-Reece U, Jongert E, Ewer KJ, Hill AVS, Jin C, Hill J, Pollard AJ, Munir Alam S, Tomaras GD, Dennison SM. A tool for evaluating heterogeneity in avidity of polyclonal antibodies. Front Immunol. 2023 Feb 16;14:1049673. doi: 10.3389/fimmu.2023.1049673. eCollection 2023. PMID 36875126
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 114460 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114460 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114460 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114460 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114460 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114460 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ad35.CS.01 Group | GSK257049 Group | Control Group
Started | 28 | 27 | 12
Completed | 26 | 25 | 12
Not Completed | 2 | 2 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Migrated | 1 | 1 | 0
Not completed — Declined challenged | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ad35.CS.01 Group | GSK257049 Group | Control Group | Total
Number analyzed (Participants) | 28 | 27 | 12 | 67
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.9 (7.03) | 30.3 (7.83) | 29.8 (6.86) | 30.04 (7.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 10 | 6 | 32
  Male | 12 | 17 | 6 | 35
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Races: African heritage/African American | 9 | 16 | 5 | 30
  Races: American Indian or Alaskan native | 0 | 1 | 0 | 1
  Races: Asian - Central/South Asian heritage | 1 | 1 | 1 | 3
  Races: White - Caucasian/European heritage | 15 | 9 | 5 | 29
  Races: Mixed Origin | 3 | 0 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Plasmodium Falciparum Parasitemia Following Sporozoite Challenge
Description: P. falciparum parasitemia was defined as a positive blood slide.
Time Frame: 28 days following sporozoite challenge (Day 105)
Population: The analyses were performed on the According-to-Protocol (ATP) cohort for Efficacy, which included all evaluable subjects who did not use any medication or blood products forbidden by the protocol, who did not report any under lying medical condition influencing immune responses, for whom efficacy data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Ad35.CS.01 Group | GSK257049 Group | Control Group
Number analyzed (Participants) | 25 | 21 | 12
Participants | 14 | 10 | 12
Statistical Analysis 1: Comparison: Ad35.CS.01 Group vs GSK257049 Group; Comparison of the efficacy (occurrence of P. falciparum parasitemia, assessed by blood slide) of an immunization regimen comprising of one dose of Ad35.CS.01 vaccine followed one month later by 2 doses of GSK257049 vaccine administered at one month intervals, with that of 3 doses of GSK257049 vaccine administered at one month intervals, in healthy malaria-naïve volunteers aged 18-50 years in the sporozoite challenge model; Test type: Other; p = 0.7675, 2-sided Fisher Exact test; Vaccine Efficacy Maentel-Haenzel Method = -17.6, 95% CI 2-sided [-107.4 to 33.3] — Pre-defined futility criteria for efficacy: point estimate of increase of VE in Ad35.CS.01 Group over GSK257049 Group less than 0%
Statistical Analysis 2: Comparison: Ad35.CS.01 Group vs Control Group; Comparison of the efficacy (occurrence of P. falciparum parasitemia, assessed by blood slide) of an immunization regimen comprising of one dose of Ad35.CS.01 vaccine followed one month later by 2 doses of GSK257049 vaccine administered at 1 month intervals, with that of 3 doses of GSK257049 vaccine administered at one month intervals, in healthy malaria-naïve volunteers aged 18-50 years in the sporozoite challenge model; Test type: Other; p = 0.0066, 2-sided Fisher Exact test; Vaccine Efficacy: Maentel-Haenzel Method = 44.0, 95% CI 2-sided [20.7 to 60.4]
Statistical Analysis 3: Comparison: GSK257049 Group vs Control Group; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.0021, 2-sided Fisher Exact test; Vaccine Efficacy: Maentel-Haenzel Method = 52.4, 95% CI 2-sided [25.4 to 69.6]

2. Primary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = significant pain at rest, pain that prevented normal every day activities. Grade 3 redness/swelling = redness/swelling spreading beyond 100 millimeters (mm) of injection site.
Time Frame: Within the 7-day (Day 0 - Day 6) follow-up period post-vaccination
Population: The analyses were performed on the Intention-to-treat (ITT) cohort, which included all subjects with at least one vaccine administration documented, who had their symptoms sheet filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | Ad35.CS.01 Group | GSK257049 Group
Number analyzed (Participants) | 28 | 27
Participants
  Any Pain, Dose 1 | 25 | 25
  Grade 3 Pain, Dose 1 | 0 | 1
  Any Redness, Dose 1 | 7 | 4
  Grade 3 Redness, Dose 1 | 0 | 0
  Any Swelling, Dose 1 | 6 | 6
  Grade 3 Swelling, Dose 1 | 0 | 0
  Any Pain, Dose 2 | 26 | 20
  Grade 3 Pain, Dose 2 | 1 | 0
  Any Redness, Dose 2 | 8 | 7
  Grade 3 Redness, Dose 2 | 1 | 0
  Any Swelling, Dose 2 | 6 | 3
  Grade 3 Swelling, Dose 2 | 0 | 0
  Any Pain, Dose 3: number analyzed (Participants) | 26 | 27
  Any Pain, Dose 3 | 20 | 15
  Grade 3 Pain, Dose 3: number analyzed (Participants) | 26 | 27
  Grade 3 Pain, Dose 3 | 1 | 0
  Any Redness, Dose 3: number analyzed (Participants) | 26 | 27
  Any Redness, Dose 3 | 11 | 8
  Grade 3 Redness, Dose 3: number analyzed (Participants) | 26 | 27
  Grade 3 Redness, Dose 3 | 0 | 1
  Any Swelling, Dose 3: number analyzed (Participants) | 26 | 27
  Any Swelling, Dose 3 | 10 | 6
  Grade 3 Swelling, Dose 3: number analyzed (Participants) | 26 | 27
  Grade 3 Swelling, Dose 3 | 0 | 0
  Any Pain, Across Doses | 27 | 26
  Grade 3 Pain, Across Doses | 2 | 1
  Any Redness, Across Doses | 15 | 11
  Grade 3 Redness, Across Doses | 1 | 1
  Any Swelling, Across Doses | 13 | 11
  Grade 3 Swelling, Across Doses | 0 | 0

3. Primary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were chills, fatigue, gastrointestinal symptoms, headache and temperature [defined as axillary temperature equal to or above (≥) 38 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade.Grade 3 Chills = rigors [uncontrollable shivering more than (>) 15 seconds]. Grade 3 Fatigue, Gastrointestinal symptoms and Headache = symptoms that prevented normal activity. Grade 3 fever = fever higher than (>) 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: Within the 7-day (Day 0 - Day 6) follow-up period post-vaccination
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Ad35.CS.01 Group | GSK257049 Group
Number analyzed (Participants) | 28 | 27
Participants
  Any Chills, Dose 1 | 7 | 3
  Related Chills, Dose 1 | 7 | 3
  Grade 3 Chills, Dose 1 | 2 | 1
  Any Fatigue, Dose 1 | 9 | 11
  Related Fatigue, Dose 1 | 9 | 8
  Grade 3 Fatigue, Dose 1 | 0 | 1
  Any Gastrointestinal symptoms, Dose 1 | 3 | 4
  Related Gastrointestinal symptoms, Dose 1 | 3 | 3
  Grade 3 Gastrointestinal symptoms, Dose 1 | 0 | 1
  Any Headache, Dose 1 | 12 | 10
  Related Headache, Dose 1 | 11 | 7
  Grade 3 Headache, Dose 1 | 0 | 2
  Any Temperature, Dose 1 | 3 | 2
  Related Temperature, Dose 1 | 2 | 2
  Grade 3 Temperature, Dose 1 | 0 | 0
  Any Chills, Dose 2 | 6 | 11
  Related Chills, Dose 2 | 6 | 11
  Grade 3 Chills, Dose 2 | 0 | 1
  Any Fatigue, Dose 2 | 9 | 11
  Related Fatigue, Dose 2 | 8 | 11
  Grade 3 Fatigue, Dose 2 | 0 | 0
  Any Gastrointestinal symptoms, Dose 2 | 0 | 1
  Related Gastrointestinal symptoms, Dose 2 | 0 | 1
  Grade 3 Gastrointestinal symptoms, Dose 2 | 0 | 0
  Any Headache, Dose 2 | 10 | 12
  Related Headache, Dose 2 | 9 | 11
  Grade 3 Headache, Dose 2 | 0 | 0
  Any Temperature, Dose 2 | 1 | 3
  Related Temperature, Dose 2 | 1 | 3
  Grade 3 Temperature, Dose 2 | 0 | 0
  Any Chills, Dose 3: number analyzed (Participants) | 26 | 27
  Any Chills, Dose 3 | 8 | 7
  Related Chills, Dose 3: number analyzed (Participants) | 26 | 27
  Related Chills, Dose 3 | 8 | 7
  Grade 3 Chills, Dose 3: number analyzed (Participants) | 26 | 27
  Grade 3 Chills, Dose 3 | 2 | 1
  Any Fatigue, Dose 3: number analyzed (Participants) | 26 | 27
  Any Fatigue, Dose 3 | 8 | 10
  Related Fatigue, Dose 3: number analyzed (Participants) | 26 | 27
  Related Fatigue, Dose 3 | 8 | 9
  Grade 3 Fatigue, Dose 3: number analyzed (Participants) | 26 | 27
  Grade 3 Fatigue, Dose 3 | 1 | 0
  Any Gastrointestinal symptoms, Dose 3: number analyzed (Participants) | 26 | 27
  Any Gastrointestinal symptoms, Dose 3 | 3 | 2
  Related Gastrointestinal symptoms, Dose 3: number analyzed (Participants) | 26 | 27
  Related Gastrointestinal symptoms, Dose 3 | 3 | 1
  Grade 3 Gastrointestinal symptoms, Dose 3: number analyzed (Participants) | 26 | 27
  Grade 3 Gastrointestinal symptoms, Dose 3 | 0 | 0
  Any Headache, Dose 3: number analyzed (Participants) | 26 | 27
  Any Headache, Dose 3 | 14 | 6
  Related Headache, Dose 3: number analyzed (Participants) | 26 | 27
  Related Headache, Dose 3 | 14 | 6
  Grade 3 Headache, Dose 3: number analyzed (Participants) | 26 | 27
  Grade 3 Headache, Dose 3 | 1 | 0
  Any Temperature, Dose 3: number analyzed (Participants) | 26 | 27
  Any Temperature, Dose 3 | 2 | 5
  Related Temperature, Dose 3: number analyzed (Participants) | 26 | 27
  Related Temperature, Dose 3 | 2 | 4
  Grade 3 Temperature, Dose 3: number analyzed (Participants) | 26 | 27
  Grade 3 Temperature, Dose 3 | 1 | 0
  Any Chills, Across doses | 15 | 13
  Related Chills, Across doses | 15 | 13
  Grade 3 Chills, Across doses | 4 | 3
  Any Fatigue, Across doses | 15 | 17
  Related Fatigue, Across doses | 15 | 14
  Grade 3 Fatigue, Across doses | 1 | 1
  Any Gastrointestinal symptoms, Across doses | 5 | 6
  Related Gastrointestinal symptoms, Across doses | 5 | 5
  Grade 3 Gastrointestinal symptoms, Across doses | 0 | 1
  Any Headache, Across doses | 21 | 14
  Related Headache, Across doses | 21 | 13
  Grade 3 Headache, Across doses | 1 | 2
  Any Temperature, Across doses | 6 | 9
  Related Temperature, Across doses | 5 | 8
  Grade 3 Temperature, Across doses | 1 | 0

4. Primary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: Within the 30-day (Day 0 - Day 29) follow-up period post-vaccination
Population: The analyses were performed on the Intention-to-treat (ITT) cohort, which included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Ad35.CS.01 Group | GSK257049 Group
Number analyzed (Participants) | 28 | 27
Participants | 23 | 21

5. Primary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs)
Description: as for outcome 4
Time Frame: Within the 30-day (Day 0 - Day 29) follow-up period post-challenge
Population: The analyses were performed on the Intention-to-treat (ITT) cohort, which included all subjects with at least one vaccine administration documented. All challenged infectivity controls were also included in this cohort and presented as a separate group.
Measure: Count of Participants; unit: Participants
Arm/Group | Ad35.CS.01 Group | GSK257049 Group | Control Group
Number analyzed (Participants) | 25 | 21 | 12
Participants | 22 | 18 | 12

6. Primary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: Throughout the study period (Day 0 - Day 236)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Ad35.CS.01 Group | GSK257049 Group | Control Group
Number analyzed (Participants) | 28 | 27 | 12
Participants | 0 | 0 | 0

7. Secondary Outcome: Number of Days Until the Onset of P. Falciparum Parasitemia Following Sporozoite Challenge
Description: The onset of P. falciparum parasitemia was defined by a positive blood slide.
Time Frame: From day of challenge (Day 0) up to 159 days post-challenge
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Ad35.CS.01 Group | GSK257049 Group | Control Group
Number analyzed (Participants) | 14 | 10 | 12
Days | 14 (1) | 14 (2) | 12 (2)

8. Secondary Outcome: Anti-circumsporozoite Protein (Anti-CS) Antibody Titers
Description: Titers are presented as geometric mean titers (GMTs) and are measured in titers. Volunteers from Control Group did not receive any immunization, but were subjected to the sporozoite challenge, therefore GMTs for this group are presented as from Day 77.
Time Frame: 28 days post-dose 1 (Day 28), 28 days post-dose 2 (Day 56), 21 days post-dose 3 (Day 77 = Day of challenge), 28 days post-challenge (Day 105), 63 days post-challenge (Day 140), 159 days post-challenge (Day 236)
Population: The analyses were performed on the According-to-Protocol (ATP) cohort for Immunogenicity, which included all evaluable subjects who met all eligibility criteria, who complied with the protocol requirements, who did not report any underlying medical condition influencing immune responses and for whom immunogenicity data were available.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Ad35.CS.01 Group | GSK257049 Group | Control Group
Number analyzed (Participants) | 26 | 27 | 12
Titers
  D28: number analyzed (Participants) | 26 | 27 | 0
  D28 | 0.9 [0.6 to 1.4] | 14.7 [8.7 to 24.9] |
  D56: number analyzed (Participants) | 26 | 27 | 0
  D56 | 14.3 [9.4 to 21.6] | 79.2 [51.0 to 122.9] |
  D77: number analyzed (Participants) | 25 | 22 | 12
  D77 | 55.5 [40.2 to 76.6] | 115.9 [77.0 to 174.5] | 0.3 [0.3 to 0.3]
  D105: number analyzed (Participants) | 25 | 21 | 12
  D105 | 50.0 [36.0 to 69.5] | 96.6 [61.3 to 152.2] | 0.5 [0.2 to 1.5]
  D140: number analyzed (Participants) | 25 | 27 | 12
  D140 | 40.5 [28.9 to 56.8] | 62.3 [42.5 to 91.2] | 0.4 [0.2 to 0.8]
  D236: number analyzed (Participants) | 26 | 25 | 12
  D236 | 21.4 [15.3 to 30.1] | 29.2 [19.7 to 43.4] | 0.3 [0.2 to 0.5]

9. Secondary Outcome: Anti-hepatitis B (Anti-HBs) Antibody Titers
Description: as for outcome 8
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Ad35.CS.01 Group | GSK257049 Group | Control Group
Number analyzed (Participants) | 26 | 27 | 12
Titers
  D28: number analyzed (Participants) | 26 | 27 | 0
  D28 | 53.0 [15.7 to 179.1] | 26596.6 [6100.1 to 115962.1] |
  D56: number analyzed (Participants) | 26 | 27 | 0
  D56 | 15845.4 [3349.8 to 74953.1] | 59388.2 [21718.8 to 162392.0] |
  D77: number analyzed (Participants) | 25 | 22 | 12
  D77 | 30877.5 [11760.6 to 81068.5] | 103746.8 [46444.1 to 231749.9] | 35.6 [5.3 to 240.6]
  D105: number analyzed (Participants) | 25 | 21 | 12
  D105 | 28180.7 [12190.4 to 65145.8] | 77659.2 [35596.0 to 169427.8] | 47.4 [7.3 to 308.9]
  D140: number analyzed (Participants) | 25 | 27 | 12
  D140 | 29307.7 [14002.8 to 61340.8] | 47932.8 [22214.7 to 103424.7] | 41.2 [6.4 to 265.8]
  D236: number analyzed (Participants) | 26 | 25 | 12
  D236 | 15589.7 [7898.8 to 30768.9] | 40727.8 [18101.6 to 91636.2] | 34.2 [6.3 to 187.1]

10. Secondary Outcome: Anti-Adenovirus Type 35 (Ad35) Neutralizing Antibody Titers at Specified Time Points
Description: as for outcome 8
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Ad35.CS.01 Group | GSK257049 Group | Control Group
Number analyzed (Participants) | 26 | 27 | 12
Titers
  D28: number analyzed (Participants) | 26 | 27 | 0
  D28 | 27.3 [17.4 to 43.0] | 16.3 [15.7 to 17.0] |
  D56: number analyzed (Participants) | 26 | 27 | 0
  D56 | 25.5 [16.6 to 39.1] | 16.5 [15.5 to 17.7] |
  D77: number analyzed (Participants) | 25 | 22 | 12
  D77 | 26.3 [16.6 to 41.5] | 17.0 [15.6 to 18.6] | 23.2 [13.3 to 40.7]
  D105: number analyzed (Participants) | 25 | 21 | 12
  D105 | 22.1 [14.6 to 33.5] | 17.2 [15.3 to 19.4] | 25.9 [13.4 to 50.0]
  D140: number analyzed (Participants) | 25 | 27 | 12
  D140 | 20.8 [14.3 to 30.1] | 16.0 [16.0 to 16.0] | 23.4 [14.2 to 38.7]
  D236: number analyzed (Participants) | 26 | 25 | 12
  D236 | 21.3 [15.5 to 29.3] | 16.5 [15.5 to 17.5] | 24.2 [14.1 to 41.5]

11. Secondary Outcome: Frequency of CS (Total CS or Repeat)-Specific CD4+ T-cells
Description: CS-specific CD4+ T-cells expressing at least 2 cytokines/activation markers between IL-2, IFN-γ, TNF-α and CD40-L are presented here. Analysis was performed via intra-cellular staining (ICS) assays, data are presented as frequency of T-cells per million peripheral blood mononuclear cells (PBMCs).Volunteers from Control Group did not receive any immunization, but were subjected to the sporozoite challenge, therefore the frequency for this group is presented as from Day 77.
Time Frame: 14 days post-dose 1 (Day 14), 14 days post-dose 2 (Day 42), 21 days post-dose 3 (Day 77 = Day of challenge), 28 days post-challenge (Day 105), 63 days post-challenge (Day 140), 159 days post-challenge (Day 236)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: T-cells/million PBMCs
Arm/Group | Ad35.CS.01 Group | GSK257049 Group | Control Group
Number analyzed (Participants) | 26 | 24 | 11
T-cells/million PBMCs
  D14: number analyzed (Participants) | 26 | 24 | 0
  D14 | 143.23 (170.19) | 220.25 (188.34) |
  D42: number analyzed (Participants) | 26 | 24 | 0
  D42 | 1693.38 (1268.50) | 854.29 (911.56) |
  D77: number analyzed (Participants) | 21 | 17 | 6
  D77 | 1364.95 (1025.92) | 608.59 (744.99) | 96.00 (94.72)
  D105: number analyzed (Participants) | 17 | 15 | 10
  D105 | 1149.29 (560.47) | 622.27 (448.50) | 80.90 (88.40)
  D140: number analyzed (Participants) | 19 | 22 | 10
  D140 | 893.68 (933.95) | 492.14 (424.34) | 36.40 (75.39)
  D236: number analyzed (Participants) | 19 | 16 | 11
  D236 | 750.95 (676.98) | 363.69 (272.73) | 59.55 (65.07)

12. Secondary Outcome: Frequency of CS (Total CS or Repeat)-Specific CD8+ T Cells
Description: CS-specific CD8+ T-cells expressing at least 2 cytokines/activation markers between IL-2, IFN-γ, TNF-α and CD40-L are presented here. Analysis was performed via intra-cellular staining (ICS) assays, data are presented as frequency of T-cells per million peripheral blood mononuclear cells (PBMC). Volunteers from Control Group did not receive any immunization, but were subjected to the sporozoite challenge, therefore the frequency for this group is presented as from Day 77.
Time Frame: as for outcome 11
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: T-cells/million PBMCs
Arm/Group | Ad35.CS.01 Group | GSK257049 Group | Control Group
Number analyzed (Participants) | 26 | 24 | 11
T-cells/million PBMCs
  D14: number analyzed (Participants) | 26 | 24 | 0
  D14 | 37.04 (64.66) | 18.29 (33.10) |
  D42: number analyzed (Participants) | 26 | 24 | 0
  D42 | 76.81 (107.06) | 25.29 (37.31) |
  D77: number analyzed (Participants) | 21 | 17 | 6
  D77 | 94.86 (153.45) | 31.35 (34.89) | 19.00 (32.21)
  D105: number analyzed (Participants) | 17 | 15 | 10
  D105 | 131.47 (153.24) | 32.27 (40.73) | 8.50 (16.43)
  D140: number analyzed (Participants) | 19 | 22 | 10
  D140 | 99.95 (159.19) | 26.18 (34.99) | 44.60 (93.49)
  D236: number analyzed (Participants) | 19 | 16 | 11
  D236 | 42.74 (47.54) | 28.00 (51.66) | 48.45 (68.98)

13. Secondary Outcome: Frequency of HBs-specific CD4+ T-cells
Description: HB-specific CD4+ T-cells expressing at least 2 cytokines/activation markers between IL-2, IFN-γ, TNF-α and CD40-L are presented here. Analysis was performed via intra-cellular staining (ICS) assays, data are presented as frequency of T-cells per million peripheral blood mononuclear cells (PBMCs). Volunteers from Control Group did not receive any immunization, but were subjected to the sporozoite challenge, therefore the frequency for this group is presented as from Day 77.
Time Frame: as for outcome 11
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: T-cells/million PBMCs
Arm/Group | Ad35.CS.01 Group | GSK257049 Group | Control Group
Number analyzed (Participants) | 25 | 25 | 11
T-cells/million PBMCs
  D14: number analyzed (Participants) | 24 | 25 | 0
  D14 | 373.67 (613.02) | 1400.80 (2449.05) |
  D42: number analyzed (Participants) | 25 | 24 | 0
  D42 | 1518.36 (1526.01) | 1836.33 (2264.88) |
  D77: number analyzed (Participants) | 22 | 18 | 8
  D77 | 1163.77 (1022.03) | 1023.58 (936.22) | 232.13 (301.75)
  D105: number analyzed (Participants) | 17 | 15 | 10
  D105 | 1265.00 (863.73) | 1310.53 (747.79) | 569.70 (489.67)
  D140: number analyzed (Participants) | 19 | 22 | 10
  D140 | 1158.47 (804.40) | 1181.00 (603.43) | 531.90 (407.21)
  D236: number analyzed (Participants) | 19 | 16 | 11
  D236 | 940.16 (564.66) | 1244.38 (833.86) | 498.36 (313.94)

14. Secondary Outcome: Frequency of CS-specific T-cells Producing IFN-γ
Description: The analysis was performed via Enzyme-Linked Immunospot (ELISPOT) full length assay. Data are presented as the number of spots per million peripheral blood mononuclear cells (PBMCs). Volunteers from Control Group did not receive any immunization, but were subjected to the sporozoite challenge, therefore the frequency for this group is presented as from Day 77.
Time Frame: as for outcome 11
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: spots/million PBMCs
Arm/Group | Ad35.CS.01 Group | GSK257049 Group | Control Group
Number analyzed (Participants) | 26 | 27 | 12
spots/million PBMCs
  D14: number analyzed (Participants) | 26 | 26 | 0
  D14 | 51.05 (61.89) | 63.20 (100.85) |
  D42: number analyzed (Participants) | 26 | 27 | 0
  D42 | 297.97 (243.24) | 54.27 (53.52) |
  D77: number analyzed (Participants) | 25 | 21 | 12
  D77 | 225.98 (161.51) | 64.54 (87.40) | 66.68 (124.31)
  D105: number analyzed (Participants) | 22 | 19 | 10
  D105 | 232.35 (175.77) | 58.04 (76.86) | 90.75 (219.50)
  D140: number analyzed (Participants) | 22 | 24 | 10
  D140 | 208.97 (125.45) | 50.77 (71.69) | 75.74 (135.72)
  D236: number analyzed (Participants) | 24 | 22 | 11
  D236 | 167.91 (153.79) | 38.85 (56.36) | 105.12 (255.20)

15. Secondary Outcome: Frequency of CS-specific T-cells Producing IFN-γ
Description: The analysis was performed via Enzyme-Linked Immunospot (ELISPOT) N-terminal assay. Data are presented as the number of spots per million peripheral blood mononuclear cells (PBMCs).
Time Frame: 14 days post-dose 1 (Day 14)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: spots/million PBMCs
Arm/Group | Ad35.CS.01 Group | GSK257049 Group
Number analyzed (Participants) | 25 | 27
spots/million PBMCs | 18.88 (19.97) | 14.57 (18.39)

ADVERSE EVENTS:
Time Frame: Solicited local/general symptoms: during the 7-day post-vaccination period (Days 0-6). Unsolicited AEs: during the 31-day post-vaccination (Days 0-30). SAEs: during the entire study period (Day 0 - Day 236).
Arm/Group | Ad35.CS.01 Group | GSK257049 Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/27 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/27 | 0/12
Other Adverse Events (participants affected / at risk) | 27/28 | 27/27 | 12/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Ad35.CS.01 Group (N=28) | GSK257049 Group (N=27) | Control Group (N=12)
Nausea (post-vaccination) (Gastrointestinal disorders) | 0 | 2 | 0/0 — Subjects from Control Group did not receive any vaccination.
Fatigue (post-vaccination) (General disorders) | 2 | 0 | 0/0 — Subjects from Control Group did not receive any vaccination.
Malaise (post-vaccination) (General disorders) | 2 | 1 | 0/0 — Subjects from Control Group did not receive any vaccination.
Pain (post-vaccination) (General disorders) | 5 | 2 | 0/0 — Subjects from Control Group did not receive any vaccination.
Nasopharyngitis (post-vaccination) (Infections and infestations) | 2 | 5 | 0/0 — Subjects from Control Group did not receive any vaccination.
Upper respiratory tract infection (post-vaccination) (Infections and infestations) | 6 | 5 | 0/0 — Subjects from Control Group did not receive any vaccination.
Arthralgia (post-vaccination) (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0/0 — Subjects from Control Group did not receive any vaccination.
Back pain (post-vaccination) (Musculoskeletal and connective tissue disorders) | 4 | 1 | 0/0 — Subjects from Control Group did not receive any vaccination.
Headache (post-vaccination) (Nervous system disorders) | 3 | 4 | 0/0 — Subjects from Control Group did not receive any vaccination.
Dysmenorrhoea (post-vaccination) (Reproductive system and breast disorders) | 3 | 1 | 0/0 — Subjects from Control Group did not receive any vaccination.
Nasal congestion (post-vaccination) (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 0/0 — Subjects from Control Group did not receive any vaccination.
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0/0 — Subjects from Control Group did not receive any vaccination.
Hyperhidrosis (post-vaccination) (Skin and subcutaneous tissue disorders) | 0 | 3 | 0/0 — Subjects from Control Group did not receive any vaccination.
Pruritus (post-vaccination) (Skin and subcutaneous tissue disorders) | 2 | 2 | 0/0 — Subjects from Control Group did not receive any vaccination.
Malaria (post-challenge) (Infections and infestations) | 14/25 | 10/21 | 12 — For the post-challenge period, 25 subjects from AD35.CS.01 Group and 21 subjects from GSK257049 Group participated in the challenge procedures and had results available.
Headache (post-challenge) (Nervous system disorders) | 5/25 | 7/21 | 2 — For the post-challenge period, 25 subjects from AD35.CS.01 Group and 21 subjects from GSK257049 Group participated in the challenge procedures and had results available.
Oropharyngeal pain(post-challenge) (Respiratory, thoracic and mediastinal disorders) | 3/25 | 0/21 | 0 — For the post-challenge period, 25 subjects from AD35.CS.01 Group and 21 subjects from GSK257049 Group participated in the challenge procedures and had results available.
Nausea (post-challenge) (Gastrointestinal disorders) | 1/25 | 2/21 | 0 — For the post-challenge period, 25 subjects from AD35.CS.01 Group and 21 subjects from GSK257049 Group participated in the challenge procedures and had results available.
Upper respiratory tract infection (post-challenge) (Infections and infestations) | 1/25 | 2/21 | 2 — For the post-challenge period, 25 subjects from AD35.CS.01 Group and 21 subjects from GSK257049 Group participated in the challenge procedures and had results available.
Pruritus (post-challenge) (Skin and subcutaneous tissue disorders) | 1/25 | 2/21 | 0 — For the post-challenge period, 25 subjects from AD35.CS.01 Group and 21 subjects from GSK257049 Group participated in the challenge procedures and had results available.
Pain- solicited local (post-vaccination) (General disorders) | 27 | 26 | 0/0 — Subjects from Control Group did not receive any vaccination.
Redness (post-vaccination) (General disorders) | 15 | 11 | 0/0 — Subjects from Control Group did not receive any vaccination.
Swelling (post-vaccination) (General disorders) | 13 | 11 | 0/0 — Subjects from Control Group did not receive any vaccination.
Chills (post-vaccination) (General disorders) | 15 | 13 | 0/0 — Subjects from Control Group did not receive any vaccination.
Fatigue (post-vaccination) (General disorders) | 15 | 17 | 0/0 — Subjects from Control Group did not receive any vaccination.
Gastrointestinal symptoms (post-vaccination) (General disorders) | 5 | 6 | 0/0 — Subjects from Control Group did not receive any vaccination.
Headache- solicited general (post-vaccination) (General disorders) | 21 | 14 | 0/0 — Subjects from Control Group did not receive any vaccination.
Temperature (post-vaccination) (General disorders) | 6 | 9 | 0/0 — Subjects from Control Group did not receive any vaccination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.